CLINICAL TRIAL: NCT02001116
Title: Improving the Quality of Paediatric Hospital Care in the Kyrgyz Republic: Evaluation of the Impact of the Intervention
Brief Title: Improving the Quality of Paediatric Hospital Care in the Kyrgyz Republic
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: WHO Collaborating Centre for Maternal and Child Health, Trieste (Other)
Collaborators: World Health Organization (Other); Scientific Center of Children RAMS (Unknown); Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Marzia Lazzerini, PhD, WHO Collaborating Centre for Maternal and Child Health, Trieste
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: WHOCCT-001
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Quality of Hospital Care for Children
Keywords: Quality of care; Hospital; Children; WHO guideline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pilot Hospitals (Experimental)
  Interventions: Other: Quality Improvement intervention
- Control Hospitals (No Intervention)

INTERVENTIONS:
Other: Quality Improvement intervention — 1. Training for local trainers and medical staff on the National Adaptation of the WHO guidelines "Pocket Book of Hospital Care for Children".
  2. Regular supporting supervision and monitoring at hospital level aimed at a sustainable improvement of the quality of the paediatric hospital care
  Arms: Pilot Hospitals

SUMMARY:
A cooperation agreement between the Ministry of Health (MOH) of Kyrgyz Republic and WHO-EURO was established, for the implementation of a WHO Project to improve the quality of pediatric care in the referral hospitals. The pilot regions selected for this intervention are the three northern regions of Thalas, Chiu and Issik-Kul Region in Kyrgyz Republic. The MOH project will be implemented at a first stage in a group of 10 pilot hospitals, randomly selected among the existing hospitals in the above cited regions. Pilot Hospitals will be compared to "control hospitals", which are the hospitals in the region not receiving the intervention, using a pre-defined set of indicators of quality of care. The results of the present evaluation on the pilot hospitals will provide data that will inform the MOH on how better to scale up this project at a national scale.

ELIGIBILITY:
Inclusion Criteria:

* The study will evaluate Quality of Care delivered to children at hospital level. This will be assessed by a direct review of patients' charts, in comparison with pre-defined standard. At the hospital level children's charts will be randomly chosen among children 2 months to 59 months, hospitalized with common diseases, such as acute respiratory diseases, diarrhoea, and fever.

Exclusion Criteria:

* Children not included in the above criteria.

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4626 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Quality of Care | 12 months
  Quality of Care will be measured using 10 pre-defined indicators
  1. Inappropriate hospitalisation (i.e. versus WHO standards)
  2. Increased risk of iatrogenic adverse effects (i.e unnecessary poly-therapy, compared to WHO standards)
  3. Unnecessary pain (i.e. unnecessary injections or other invasive procedures, as compared to WHO standards)
  4. Incorrect Diagnosis (i.e. versus WHO standards)
  5. Incorrect Treatment (i.e. versus WHO standards)
  6. Inconsistency between diagnosis and treatment (i.e. versus WHO standards)
  7. Inadequate Monitoring: (i.e. versus WHO standards)
  8. Lack of nutritional evaluation (i.e. versus WHO standards)
  9. Incorrect use of IV fluids (i.e. versus WHO standards)
Primary outcome | 12 months
  Children with concomitant presence of all the following three indicators of case management: 1) unnecessary hospitalization; 2) increased risk of iatrogenic adverse effects; 3) unnecessary painful procedures

SECONDARY OUTCOMES:
Outcomes of QoC | 12 months
  Summary scores according to the WHO Quality Asessment Tool

CONTACTS AND LOCATIONS:
Locations (1):
- Thalas, Chiu and Issik-Kul Regions, Thalas, Chiu, Issik-Kul, Kyrgyzstan